CLINICAL TRIAL: NCT04383483
Title: CoV-ICU Score: Who Will Need Intensive Care in the Course of Corona Virus Disease?
Brief Title: CoV-ICU Score, Intensive Care Unit, SARS-CoV-2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Ali ASAN, Associate professor, Bursa Yuksek Ihtisas Training and Research Hospital
Other Study IDs: BYIEAH-202005
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Coronavirus as the Cause of Diseases Classified Elsewhere
Keywords: SARS-CoV-2, intensive care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CoVID patients admitted to ICU: Patients admitted to the intensive care unit with the diagnosis of COVID
  Interventions: Other: COVICU

INTERVENTIONS:
Other: COVICU — COVICU

SUMMARY:
In the course of COVID disease, some patients need intensive care treatment. We aim to find an answer to the question of whether the patient's CRP, ferritin, D-dimer, Oxygen Saturation, lymphocyte count, and body mass index can be used as a criterion for admitting patients with COVID to the intensive see unit.

DETAILED DESCRIPTION:
It is aimed to determine the patients who are above the threshold value to be determined according to this scoring result. Identifying patients who may need intensive care and following them closely will positively affect patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to the intensive care unit with the diagnosis of COVID

Exclusion Criteria:

<18 years patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the intensive care unit with the diagnosis of COVID
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
COVICU score | 1 week
  With this scoring, identifying patients who may need intensive care early and following them closely will have a positive effect on patient prognosis.
Values | 1 week
  Minimum and maximum values will be determined at the end of the study. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Ali Asan, MD, Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yüksek Ihtisas Training and Research Hospital, Bursa, Yildirim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol